CLINICAL TRIAL: NCT03047720
Title: Scheduled Awakenings for the Treatment of Nocturnal Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Benjamin Whittam, Assistant Professor of Urology, Indiana University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1601620278
Record Dates: First submitted 2016-12-28; First posted 2017-02-09 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Nocturnal Enuresis
Keywords: bedwetting
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- One: Study Phases (S1 and S2) (Other): The therapeutic phase of this study for the participant in Arm One will be: 6 weeks of behavioral modifications plus the Lully device (S1), followed by 6 weeks of behavioral modifications only without the device (S2)
  Interventions: Device: Lully Sleep Guardian
- Two: Study Phases (S2 and S1) (Other): The therapeutic phase of this study for the participant in Arm Two will be: 6 weeks of behavioral modifications only without the device (S2), followed by 6 weeks of behavioral modifications plus use of the Lully device(S1)
  Interventions: Device: Lully Sleep Guardian

INTERVENTIONS:
Device: Lully Sleep Guardian — In the initial phase, participant baseline is established. In the Therapeutic Phase, each participant will complete the study phases (S1 and S2) in the order determined by their assigned treatment arm. During the scheduled awakening protocol using Lully Sleep Guardian, a scheduled awakening will be performed each night with the Lully pod.
  During the initial and therapeutic phases of this study, participants are asked to enter responses daily into a Lully Study app. The app will send a prompt each morning. The questions the participant is prompted to answer serve to document occurrence of bedwetting and the degree of wetness.
  In addition, the family will complete the KIDSCREEN 27 and the Vancouver questionnaire at defined intervals throughout the study.
  Arms: One: Study Phases (S1 and S2)
Device: Lully Sleep Guardian — In the initial phase, participant baseline is established. In the Therapeutic Phase, each participant will complete the study phases (S1 and S2) in the order determined by their assigned treatment arm. During the scheduled awakening protocol using Lully Sleep Guardian, a scheduled awakening will be performed each night with the Lully pod.
  During the initial and therapeutic phases of this study, participants are asked to enter responses daily into a Lully Study app. The app will send a prompt each morning. The questions the participant is prompted to answer serve to document occurrence of bedwetting and the degree of wetness.
  In addition, the family will complete the KIDSCREEN 27 and the Vancouver questionnaire at defined intervals throughout the study.
  Arms: Two: Study Phases (S2 and S1)

SUMMARY:
This study is a simple effectiveness trial to determine if the Lully Sleep Guardian has any effect on benign nocturnal enuresis.

DETAILED DESCRIPTION:
Primary monosymptomatic nocturnal enuresis (PMNE) is defined by the Diagnostic & Statistical Manual of Mental Disorders (DSM- IV) as an involuntary voiding of urine during sleep, with a severity of at least twice a week, in children aged >5 years in the absence of congenital or acquired defects of the central nervous system(1-3).

PMNE affects 10-20% kids at 5 years old (1, 4, 5). It does resolve spontaneously so that 5% of 10 year olds and 1% of 15 year olds are still affected (2-4). Is more common in boys. While the disease its self is benign, and improves without intervention, it does pose a significant social and emotional burden on the child and their family. These include parental disapproval, sibling teasing, and inability to attend sleep overs with peers, all of which lead to families seeking treatment options (3, 4).

Current treatments start with conservative management. This includes appropriate fluid intake, scheduled toileting during the day, avoidance of bladder irritants and constipation (4, 5). If these fail to improve symptoms or families are looking for a more active form of treatment, first line therapy is either a bed wetting alarms or desmopressin (1, 4, 5).

The Lully Sleep Guardian was initially developed for use in night terrors. The device works by programing a vibrating disk that is placed under the child's bed to alter sleep patterns and prevent the onset of sleep terrors. The child is not woken up for the treatment of sleep terrors. The device has also been shown to anecdotally improve users' nocturnal enuresis. There have been no reports of safety concerns or hazards with the device (7, 8).

The aim of this study is to determine the effectiveness of scheduled awakenings, with the Lully Sleep Guardian, in patients with PMNE, at reducing the frequency of bed-wetting.

ELIGIBILITY:
Inclusion Criteria:

* Benign nocturnal enuresis
* Age: 5 - 17
* Must have or have access to an Apple iPhone, iPad, or iPod Touch

Exclusion Criteria:

* Diurnal Enuresis
* Constipation
* Neurogenic Bladder
* Any serious underlying cardiopulmonary problems that require diuretics or antihypertensive medications to manage
* Any bladder active medications
* Age: < 5 years of age; > 17 years of age
* Cerebral Palsy
* Mental disorders, mood disorders, or autism-spectrum disorder
* Epilepsy or seizure history
* Restless leg syndrome
* Use of benzodiazepine/clonidine

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Whittam, MD, Principal Investigator — Pediatric Urology, Riley Children's Hospital
Locations (1):
- Riley Hopspital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] National Clinical Guideline Centre (UK). Nocturnal Enuresis: The Management of Bedwetting in Children and Young People. London: Royal College of Physicians (UK); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK62712/ PMID 22031959
- [Background] Ahmed AF, Amin MM, Ali MM, Shalaby EA. Efficacy of an enuresis alarm, desmopressin, and combination therapy in the treatment of saudi children with primary monosymptomatic nocturnal enuresis. Korean J Urol. 2013 Nov;54(11):783-90. doi: 10.4111/kju.2013.54.11.783. Epub 2013 Nov 6. PMID 24255762
- [Background] Glazener CM, Evans JH, Peto RE. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2003;(2):CD002911. doi: 10.1002/14651858.CD002911. PMID 12804443
- [Background] Bayne AP, Skoog SJ. Nocturnal enuresis: an approach to assessment and treatment. Pediatr Rev. 2014 Aug;35(8):327-34; quiz 335. doi: 10.1542/pir.35-8-327. PMID 25086164
- [Background] Monda JM, Husmann DA. Primary nocturnal enuresis: a comparison among observation, imipramine, desmopressin acetate and bed-wetting alarm systems. J Urol. 1995 Aug;154(2 Pt 2):745-8. PMID 7609169
- [Background] Onol FF, Guzel R, Tahra A, Kaya C, Boylu U. Comparison of long-term efficacy of desmopressin lyophilisate and enuretic alarm for monosymptomatic enuresis and assessment of predictive factors for success: a randomized prospective trial. J Urol. 2015 Feb;193(2):655-61. doi: 10.1016/j.juro.2014.08.088. Epub 2014 Aug 23. PMID 25158273
- [Background] 7.Rink A. Lully Sleep Guardian. In: Heinsimer K, editor. IU Health2016.
- [Background] 8. Lully Sleep Guardian - Proven to Stop Night Terrors: Amazon; 2016 [cited 2015 2016]. Available from: http://www.amazon.com/Lully-Sleep-Guardian-Proven-Terrors/dp/B011LOUNCI/ref=sr_1_1?ie=UTF8&qid=1457660065&sr=8-1-spons&keywords=lully+sleep+guardian&psc=1#customerReviews.

RESULTS

PARTICIPANT FLOW:
Groups:
- Lully Device First, Then No Device: Lully device plus Behavioral modifications plus for daily for 6 weeks (S1), followed behavioral modifications only without the device daily for 6week (S2)
  No washout period between S1 and S2 because there was no carryover effect from either intervention
- No Device First, Then Lully Device: Behavioral modifications only without the device (S2) daily for 6weeks, followed by of behavioral modifications plus use of the Lully device daily for 6 weeks(S1)
  No washout period between S2 and S1 because there was no carryover effect from either intervention
Period: First Intervention (6weeks)
Arm/Group | Lully Device First, Then No Device | No Device First, Then Lully Device
Started | 12 | 0
Completed | 5 | 0
Not Completed | 7 | 0
Not completed — Participant data entry insufficient | 7 | 0
Period: Second Intervention (6weeks)
Arm/Group | Lully Device First, Then No Device | No Device First, Then Lully Device
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants did not show continued desire to document daily data after ending study phase one and discontinuing use of the Lully device
Groups:
- Total: Total of all reporting groups
Arm/Group | Lully Device First, Then No Device | No Device First, Then Lully Device | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 |  | 12
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 6 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 11 |  | 11
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Vancouver Questionnaire Score [Mean (Standard Deviation); unit: units on a scale] — The Vancouver is a 14 item questionnaire for diagnosing Dysfunctional Elimination Syndrome (DES). There is a 5-point Likert scale used for all questions. Item score range from 0 (no complaint) to 4 (severe symptoms). Question 1-13 probe for a single symptom. Question 14 speaks to ease of completing the questions. For this study, subjects with a Vancouver score less < or = to 11 (for questions 1-13) met the criteria for benign nocturnal enuresis and were determined eligible to participate. Score > 11 met criteria for DES. Total score range (for 1-13): min score of 0 to max of 52.
  units on a scale | 9.28 (3.10) |  | 9.28 (3.10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Dry Nights When Using the Scheduled Awakening Protocol With the Lully Sleep Guardian
Description: Participants were asked to enter responses daily into a Lully Study app.The questions the participant was prompted to answer: Did your child have a bed wetting episode last night? Answered by yes or no.
Time Frame: baseline and 6 weeks (end of S1)
Population: Participants who completed at least 37 nights of data entry using the scheduled awakening protocol with the Lully Sleep Guardian
Measure: Mean (Full Range); unit: difference in number of dry nights
Groups:
- Lully Device: Participants who completed 6 weeks of behavioral modifications plus the Lully device
- No Device: Participants who completed 6 weeks of behavioral modifications only without the device
Arm/Group | Lully Device | No Device
Number analyzed (Participants) | 5 | 0
difference in number of dry nights | -0.67 [-3 to 2] |

2. Primary Outcome: Change in Number of Voids Per Night When Using the Scheduled Awakening Protocol With the Lully Sleep Guardian
Description: Participants were asked to enter responses daily into a Lully Study app.The questions the participant was prompted to answer: Did your child have a bed wetting episode last night? (Answered by yes or no) What time?
Time Frame: Not measured.
Population: Unable to measure because data was not collected.
Arm/Group | Lully Device | No Device
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Quantity of Wetness When Bedwetting Occurred While Using the Scheduled Awakening Protocol With the Lully
Description: Participants were asked to enter responses daily into a Lully Study app. In a free text box the family was asked to add additional information to describe how wet the child was using the following 1-5 scale: 1- wet underwear; 2-wet underwear and damp pajamas; 3- soaked underwear, pajamas; 4-soaked pajamas, damp mattress; 5- soaked mattress.
Time Frame: Not measured.
Population: No participant were analyzed. Data was not available. Contributors: data not entered by participants and app glitches could have lead to lost data if entered
Arm/Group | Lully Device | No Device
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: QOL Measures Using the KIDS Screen Questionnaire at 10 Weeks
Description: Participants were asked to complete QOL survey (KIDSCREEN 27) at baseline, before starting therapeutic phase, and after completing therapeutic phase. KIDSCREEN is a standardized questionnaire for children and adolescents to assess their health related quality of life (HRQoL). Each items scored on a 5-point scale. There is the KIDSCREEN 54 (long version) KIDSCREEN 27 (short version) KIDSCREEN 10 Index. For analysis, decision made to analyze questions in the KIDSCREEN 10 Index questions only. For KIDSCREEN 10, it is a 5 point Likert Scale with a score range of 10 to 50 with higher scores indicating better quality of life.
Time Frame: 10 weeks
Population: Patients analyzed completed the KIDSCREEN after completing the 6 weeks use of the Lully device. 4 of 5 who completed the 6 weeks use the Lully device completed the KIDSCREEN. Data was not collected for Baseline and 4 wk scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lully Device | No Device
Number analyzed (Participants) | 4 | 0
score on a scale | 42.75 (5.97) |

ADVERSE EVENTS:
Time Frame: 6weeks
Description: The number of participants in ARM 2 at risk all-cause mortality, SAEs, and other adverse events was zero because no patients advanced to that arm.
Groups:
- S1: Lully Device Plus Behavioral Modifications: The S1 therapeutic phase of this study was: 6 weeks of behavioral modifications plus the Lully device
  The family received counseling on behavioral modifications during initial baseline phase to follow throughout S1.
  During this phase, a scheduled awakening was performed each night with the Lully pod following the scheduled awakening protocol using Lully Sleep Guardian. This was used to reliably produce a brief awakening by titrating the device to a minimal awakening stimulus during the first night of use. If the brief awakening could not be produced using the Lully pod, the parent was to gently awaken the child
  Participants were asked to enter responses daily into a Lully Study app. The questions the participant was prompted to answer were to serve to document occurrence of bedwetting and the degree of wetness.
  In addition, the family were asked to complete the KIDSCREEN 27 and the Vancouver questionnaire at defined intervals
- S2: Behavioral Modifications Only: The S2 therapeutic phase of this study : 6 weeks of behavioral modifications only without the device.
  The family received counseling on behavioral modifications during initial baseline phase to follow throughout S1.
  During this phase, participants were asked to enter responses daily into a Lully Study app. The questions the participant was prompted to answer were to serve to document occurrence of bedwetting and the degree of wetness.
  In addition, the family were asked to complete the KIDSCREEN 27 and the Vancouver questionnaire at defined intervals
Arm/Group | S1: Lully Device Plus Behavioral Modifications | S2: Behavioral Modifications Only
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0

LIMITATIONS AND CAVEATS:
Study N too small to perform statistical analysis. Limits included decreased bedwetting during baseline, inconsistent user data entry in app, app glitches, lack of participant interest in proceeding to S2 after completing S1. Study ended early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT03047720/ICF_000.pdf
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03047720/Prot_001.pdf